CLINICAL TRIAL: NCT05044286
Title: An Observational Study to Understand Acceptability of Long-Acting Pre-Exposure Prophylaxis for HIV-1 Prevention in Transgender and Gender Diverse Populations in Texas
Brief Title: Longer-Acting PrEP in Transgender and Gender Diverse Texans
Status: Completed | Type: Observational
Sponsor: University of Texas at Austin (Other)
Collaborators: Texas Health Institute (Unknown); Merck Sharp & Dohme LLC (Industry); Transgender Education Network of Texas (Unknown)
Responsible Party: Principal Investigator, Phillip Schnarrs, Associate Professor, University of Texas at Austin
Other Study IDs: MISP# 60761
Record Dates: First submitted 2021-09-01; First posted 2021-09-14 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: HIV-1-infection
Keywords: Transgender; Gender Diverse; Longer-acting pre-exposure prophylaxis (PrEP); Biomedical HIV prevention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 40 Transgender and Gender Diverse for World Café Conversation: We will host two world cafe conversations. The first (n = 20) will be specifically or black transgender and gender diverse adults (18+), who are HIV-negative, and have indications for PrEP. The second (n = 20) will be open to transgender and gender diverse adults, who are HIV-negative, and have indication for PrEP.
  Interventions: Other: no intervention
- 20 Other Key stakeholders for World Café Conversation: We will interview 20 other key stakeholders including medical providers, HIV prevention specialists, outreach workers, PrEP navigators/educators.
  Interventions: Other: no intervention
- 500 Transgender and Gender Diverse for Survey: We will survey 500 TGD adults (18+), who are HIV negative, and have indications for PrEP.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The long-term goal of this project is to increase uptake and adherence of LA-PrEP in TGD populations in Texas. The central hypothesis is that strategies to increase uptake of LA- PrEP that are patient centered and understand the needs of TGD people will improve uptake and adherence. The objective of this observational study is to investigate barriers, facilitators, and preferences regarding willingness and intention to use LA-PrEP in TGD populations in Texas. Data from this study will support future research on patient centered strategies for uptake and adherence of LA-PrEP in TGD populations.

DETAILED DESCRIPTION:
Pre-exposure prophylaxis (PrEP) is a biomedical HIV prevention strategy that is more than 90% effective in preventing the transmission of HIV. Despite the promise of PrEP in eradicating HIV, uptake has been slow in transgender and gender diverse (TGD) individuals with only 3% of TGD individuals using PrEP. While awareness is a key factor related to PrEP uptake, TGD experience numerous contextual and structural barriers, including discrimination and mistreatment by medical providers, lack of availability and access (e.g., insurance, transportation, time), and broad distrust of the healthcare system that affect intention to use PrEP and reduce uptake. These barriers are further compounded by the social position of TGD people on which they are further stratified based on their race, ethnicity, and socioeconomic status. In addition to contextual and structural factors there are a number of individual factors that limit uptake including fear of side effects, issues with adherence, concerns related to stigma, and lack of trust in the medication's efficacy.

Longer-acting PrEP (LA-PrEP) regimens include different delivery modalities (e.g.. injectable, oral, subdermal implant) with different dosing protocols (e.g. monthly versus daily). There is potential for long-acting biomedical HIV prevention methods to address some of these barriers experienced by TGD individuals. However, to be successful an understanding of attitudes, norms, and other factors influencing LA-PrEP uptake and adherence is needed, specifically among racial and ethnic minority TGD individuals, and their preferences for LA-PrEP delivery. Developing patient-centered strategies for uptake and adherence, using human centered design principles will support uptake and adherence of LA-PrEP in these TGD people.

The investigators will achieve the study objective through the following aims:

Specific Aim 1. Identify factors that influence uptake and adherence of LA- PrEP among TGD individuals in Texas Activities: In collaboration with Transgender Education Network of Texas (TENT) and TransFORWARD: Texas Transgender Health (co-Is), a PCORI funded project in Texas to increase TGD patient-centered outcomes research and comparative effectiveness research capacity in Texas, the research team will recruit 40 TGD individuals to participate in a world café conversation to understand beliefs, attitudes, and preferences for LA-PrEP and interview 20 other relevant key stakeholders (e.g., medical providers, AIDS Service Organizations, TGD advocacy groups) to understand perceived barriers, facilitators, and needs regarding uptake and adherence to LA-PrEP in TGD communities. Anticipated outcomes: understanding of factors influencing uptake and adherence of LA-PrEP that will inform development of data collection instruments and provide insight about factors affecting potential LA-PrEP uptake.

Specific Aim 2: Understand factors influencing willingness and intention to use different regimens of LA- PrEP among TGD individuals living in Texas. Activities: The investigators will survey at least 500 TGD individuals from across the state about their attitudes, community norms, barriers and preferences regarding different PrEP modalities and regimens to better understand how these factors influence willingness and intention to use different forms of LA-PrEP. Anticipated Outcomes: Identification of factors that promote willingness and intention to use LA-PrEP.

ELIGIBILITY:
Inclusion Criteria: Transgender/Gender diverse, HIV negative, 18 years of age or older, Indications for PrEP, Texas resident.

Exclusion Criteria:

* HIV positive,

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Transgender and gender diverse adults living in Texas.
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Willingness to use intramuscular injectable PrEP | Data will be collected over a six month period using a cross-sectional online survey.
  Participants will be asked how willing they are to use intramuscular injectable PrEP using a 6-point Likert scale ranging from "I would definitely not use intramuscular injectable PrEP" to I would definitely use intramuscular injectable PrEP."
Willingness to use a montly oral PrEP | Data will be collected over a six month period using a cross-sectional online survey.
  Participants will be asked how willing they are to use intramuscular injectable PrEP using a 6-point Likert scale ranging from "I would definitely not use monthly oral PrEP" to I would definitely use monthly oral PrEP."
Willingness to use a yearly subdermal PrEP implant | Data will be collected over a six month period using a cross-sectional online survey.
  Participants will be asked how willing they are to use a yearly subdermal PrEP implant using a 6-point Likert scale ranging from "I would definitely not use a yearly subdermal PrEP implant" to "I would definitely use a yearly subdermal PrEP implant."

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schnarrs PW, Zuniga J, Benitez G, Fliedner P, Norwood A, Croll M, Oviedo LDS, Buchorn J, Oeffinger J, Lane R, Schelling E, Pham G, Pate T, Arnold EM. Intention to Use Different Formulations of Longer Acting HIV Pre-Exposure Prophylaxis Among Transgender and Gender Expansive Individuals: The Roles of Social Vulnerability and Medical Mistrust. AIDS Patient Care STDS. 2024 Feb;38(2):51-60. doi: 10.1089/apc.2023.0211. PMID 38381948